CLINICAL TRIAL: NCT01697488
Title: Non-interventional Surveillance Study (NIS) on First-line (FL) Bevacizumab (Avastin) in Combination With Carboplatin/Paclitaxel in Patients With Advanced Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: An Observational Study of Avastin (Bevacizumab) in Combination With Carboplatin/Paclitaxel in First Line in Patients With Advanced Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer (OTILIA)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27765
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Peritoneal Neoplasms
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort: Overall sample
- Subgroup: Patients aged >/= 70 years

SUMMARY:
This observational study will evaluate the safety, efficacy, quality of life and predictive/selection factors for Avastin (bevacizumab) in combination with carboplatin/paclitaxel in first line in patients with advanced epithelial ovarian, fallopian tube or primary peritoneal cancer in clinical practice. Data of eligible patients will be collected during up to 15 months of treatment and 12 months of follow-up. A second recruitment phase has been opened to focus on patients >/= 70 years.

ELIGIBILITY:
Inclusion Criteria:

* Study phase 1: Patients aged >/= 18 years
* Study phase 2: Patients aged >/= 70 years
* Newly diagnosed advanced epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal cancer with indication for a first-line carboplatin/paclitaxel chemotherapy in combination with Avastin

Exclusion Criteria:

* Contraindications to Avastin according to Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed advanced epithelial ovarian, fallopian tube or primary peritoneal cancer with indication for first-line carboplatin/paclitaxel chemotherapy in combination with Avastin. In the second study phase recruitment focusses on patients >/= 70 years.
Sampling Method: Probability Sample
Enrollment: 1090 (Actual)
Dates: Start 2012-02-02 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Efficacy: Progression-free survival | up to approximately 27 months
Safety: Incidence of adverse events | approximately 5 years

SECONDARY OUTCOMES:
Quality of life: European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30/QLQ-OV28 questionnaires | up to approximately 27 months
Selection criteria for first-line treatment with Avastin and carboplatin/paclitaxel: clinical/demographic patient characteristics | approximately 5 years
Treatment discontinuations/modifications | approximately 5 years
Treatment duration | approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Ortenau Klinikum Offenburg; Med. Klinik II; Mammachirurgie und Gynäkologisch-Onkologische Chirurgie, Offenburg, Germany

REFERENCES:
- [Derived] Sehouli J, Mustea A, Oskay-Ozcelik G, Keller M, Richter R, Tome O, Woopen H, Sommer-Joos AK, Grabowski JP, Armbrust R, Wimberger P. Bevacizumab Combined with Platinum-Taxane Chemotherapy as First-Line Treatment for Advanced Ovarian Cancer: Results of the NOGGO Non-Interventional Study (OTILIA) in 824 Patients. Cancers (Basel). 2021 Sep 22;13(19):4739. doi: 10.3390/cancers13194739. PMID 34638225